CLINICAL TRIAL: NCT06200168
Title: A Study on Electroacupuncture Combined With Olanzapine-contained Four-drug Antiemetic Therapy for the Prevention of Highly Emetogenic Chemotherapy-induced Nausea and Vomiting in Patients With Breast Cancer (ECO Study)
Brief Title: Electroacupuncture for the Prevention of Chemotherapy-induced Nausea and Vomiting in Patients With Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiuda Zhao (Other)
Responsible Party: Sponsor-Investigator, Jiuda Zhao, Breast Disease Diagnosis and Treatment Center, Affiliated Hospital of Qinghai University
Organization: Affiliated Hospital of Qinghai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHQU-2023002
Record Dates: First submitted 2023-12-20; First posted 2024-01-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Electroacupuncture; Olanzapine-contained Four-drug Antiemetic; Nausea and Vomiting
Keywords: electroacupuncture; olanzapine-contained four-drug antiemetic; nausea and Vomiting; breast cancer; chemotherapy
MeSH Terms: conditions — Nausea; Vomiting; Breast Neoplasms | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- True acupuncture + standard quadruple antiemetic therapy (Experimental): Participants will receive electroacupuncture once daily from day 1 to day 4. The acupuncturists will insert needles into the acupoints and manipulate the needles until"de qi"sensation is achieved and reported by the participants. Electrical stimulation will be delivered for 30 minutes at alternating frequencies of 2/10Hz. They will receive olanzapine 2.5 mg per day orally on days 1 through 4 + fosaprepitant 150 mg intravenous (IV) or aprepitant injectable emulsion 130 mg IV + palonosetron 0.25 mg IV or ondansetron 8 mg IV or tropisetron 5 mg IV (the previously mentioned medication, which includes fosaprepitant or aprepitant combined with palonosetron or ondansetron or tropisetron, can also be taken orally in a fixed combination of netupitant (300 mg) and palonosetron (0.50 mg))+ dexamethasone 10 mg IV 30 minutes prior to chemotherapy on Day 1, dexamethasone 8 mg IV on days 2, 3, 4 post chemotherapy. Dexamethasone doses may be individualized based on the doctor's judgment.
  Interventions: Device: Electroacupuncture; Drug: Standard antiemetic treatment
- Sham acupuncture + standard quadruple antiemetic therapy (Placebo Comparator): The sham acupuncture comprised a core standardized prescription of minimally invasive, shallow needle insertion using thin and short needles at body locations not recognized as true acupuncture points and are deemed to not belong to traditional Chinese meridians and have no therapeutic value. Participants will receive minimal acupuncture treatment without electrical stimulation at the same time as the intervention group.Care was taken to avoid "de qi" sensation. They will receive olanzapine-contained four-drug antiemetic therapy. All the antiemetic drugs used are the same as those in the true acupuncture group.
  Interventions: Device: Sham electroacupuncture; Drug: Standard antiemetic treatment

INTERVENTIONS:
Device: Electroacupuncture — The acupuncturists will insert needles into the acupoints and manipulate the needles until"de qi"sensation is achieved and reported by the participants. Electrical stimulation will be delivered for 30 minutes at alternating frequencies of 2/10Hz.
  Arms: True acupuncture + standard quadruple antiemetic therapy
Drug: Standard antiemetic treatment — Olanzapine 2.5 mg per day orally on days 1 through 4 + fosaprepitant 150 mg intravenous (IV) or aprepitant injectable emulsion 130 mg IV + palonosetron 0.25 mg IV or ondansetron 8 mg IV or tropisetron 5 mg IV (the previously mentioned medication, which includes fosaprepitant or aprepitant combined with palonosetron or ondansetron or tropisetron, can also be taken orally in a fixed combination of netupitant (300 mg) and palonosetron (0.50 mg))+ dexamethasone 10 mg IV 30 minutes prior to chemotherapy on Day 1, dexamethasone 8 mg IV on days 2, 3, 4 post chemotherapy. Dexamethasone doses may be individualized based on the doctor's judgment.
  Arms: True acupuncture + standard quadruple antiemetic therapy
Device: Sham electroacupuncture — The sham acupuncture comprised a core standardized prescription of minimally invasive, shallow needle insertion using thin and short needles at body locations not recognized as true acupuncture points and are deemed to not belong to traditional Chinese meridians and have no therapeutic value. Participants will receive minimal acupuncture treatment without electrical stimulation at the same time as the intervention group.Care was taken to avoid "de qi" sensation.
  Arms: Sham acupuncture + standard quadruple antiemetic therapy
Drug: Standard antiemetic treatment — Olanzapine 2.5 mg per day orally on days 1 through 4 + fosaprepitant 150 mg intravenous (IV) or aprepitant injectable emulsion 130 mg IV + palonosetron 0.25 mg IV or ondansetron 8 mg IV or tropisetron 5 mg IV (the previously mentioned medication, which includes fosaprepitant or aprepitant combined with palonosetron or ondansetron or tropisetron, can also be taken orally in a fixed combination of netupitant (300 mg) and palonosetron (0.50 mg))+ dexamethasone 10 mg IV 30 minutes prior to chemotherapy on Day 1, dexamethasone 8 mg IV on days 2, 3, 4 post chemotherapy. Dexamethasone doses may be individualized based on the doctor's judgment.All the antiemetic drugs used are the same as those in the true acupuncture group.
  Arms: Sham acupuncture + standard quadruple antiemetic therapy

SUMMARY:
This randomized controlled phase III trial aims to evaluate the use of electroacupuncture in combination with olanzapine-containing standard quadruple antiemetic drugs for the treatment of nausea and vomiting induced by highly emetogenic chemotherapy (HEC) in patients with breast cancer. Furthermore, it will analyze the relationship between single nucleotide polymorphism and electroacupuncture treatment for chemotherapy-induced nausea and vomiting.

DETAILED DESCRIPTION:
This study is a parallel-group, blinded (participants, evaluators, and statisticians), randomized controlled trial exploring the effectiveness of electroacupuncture combined with standard quadruple antiemetic drugs for breast cancer patients undergoing HEC. Both groups will receive Olanzapine, Neurokinin-1 receptor antagonists (NK-1RAs), serotonin receptor antagonists [5HT3RA], and dexamethasone at the start of HEC on Day 1. Electroacupuncture or sham acupuncture will be randomly administered to each group. Participants will document all instances of nausea and vomiting and note the use of rescue antiemetic medications. Blood samples will be collected and analyzed to investigate whether genetic polymorphisms can predict electroacupuncture outcomes in breast cancer patients undergoing HEC. Primary and secondary outcomes as well as adverse events will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older and aged 75 years or younger, of any nationality;
2. Eastern Cooperative Oncology Group performance status of 0-2;
3. Patients with breast cancer, with no restrictions on molecular typing; early-stage patients must not have undergone prior chemotherapy, while advanced-stage patients must be candidates for first-line chemotherapy and have declined neoadjuvant or adjuvant chemotherapy for over 3 months. All patients must receive highly emetogenic chemotherapy (HEC) based on anthracycline chemotherapy with cyclophosphamide (EC or AC) or carboplatin (AUC≥4)/cisplatin;
4. Predicted life expectancy of ≥3 months;
5. Adequate bone marrow, kidney, and liver function;
6. Adequate contraception if premenopausal women;
7. Written informed consent by the patient before enrolment.

Exclusion Criteria:

1. Patients already submitted to chemotherapy;
2. Is scheduled to receive any non-HEC on Day 1;
3. Is scheduled to receive any chemotherapy on days 2-4 after HEC;
4. Received or is scheduled to receive radiation therapy to the abdomen, pelvis, head and neck within 1 week prior to Day 1 or between Days 1 to 5 in cycle 1;
5. Has symptomatic primary or metastatic symptomatic central nervous system malignancy causing nausea and/or vomiting;
6. Have ongoing emesis or CTCAE grade 2 or greater nausea;
7. Significant medical or mental conditions;
8. Any allergies to study drug, antiemetics or dexamethasone;
9. Significantly abnormal laboratory values (platelets, coagulation indexes, absolute neutrophils, AST, ALT, bilirubin or creatinine);
10. Patients who are pregnant or breast-feeding;
11. Inflammatory skin reaction;
12. Has lymphedema in acupuncture stimulation area;
13. Patients who are afraid of electroacupuncture stimulation or allergic to stainless steel needles;
14. Received acupuncture treatments for any conditions less than 4 weeks before HEC;
15. Currently using drugs with antiemetic activity (e.g., 5-HT3 receptor antagonists, corticosteroids (except when used at physiological doses), dopamine receptor antagonists, minor tranquilizers, antihistamines, and benzodiazepines (except for nocturnal sedation));
16. Patients with concomitant severe diseases or with a predisposition to emesis such as gastrointestinal obstruction, active peptic ulcer, and hypercalcemia and symptomatic brain metastasis;
17. Has a convulsive disorder requiring anticonvulsant treatment;
18. Patients administered thioridazine as a chronic antipsychotic medication (patients are allowed to receive prochlorperazine and other phenothiazines as a rescue antiemetic treatment);
19. Concurrent treatment with quinolone antibiotics;
20. Has a history of chronic alcoholism (determined by the investigator);
21. Known arrhythmias, uncontrolled congestive heart failure, or acute myocardial infarction within the past six months;
22. Has a history of uncontrolled diabetes (e.g., using insulin or oral hypoglycemic agents).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with no nausea during the overall stage | 120 hours
  The proportion of patients achieving no nausea is defined as patients who have a response of 0 on the Visual Analog Scale for nausea during the overall stage (0 to 120 hours) after the initiation of chemotherapy.

SECONDARY OUTCOMES:
Proportion of patients with no nausea during the early stage | 24 hours
  The proportion of patients achieving no nausea is defined as patients who have a response of 0 on the Visual Analog Scale for nausea during the early stage (0 to 24 hours) after the initiation of chemotherapy
Proportion of patients with no nausea during the delayed stage | 96 hours
  The proportion of patients achieving no nausea is defined as patients who have a response of 0 on the Visual Analog Scale for nausea during the later stage (25 to 120 hours) after the initiation of chemotherapy
The relationship between single nucleotide polymorphism genotypes and the proportion of patients with no nausea | 120 hours
  The single nucleotide polymorphism (SNP) genotypes will be analyzed by detecting different bases (A, T, C, and G) in peripheral blood DNA. The proportion of patients with different SNP genotypes will be analyzed. The proportion of patients achieving no nausea is defined as patients who score 0 on the nausea Visual Analog Scale during the entire period (0 to 120 hours) following the initiation of chemotherapy. We will analyze the relationship between the proportion of patients with different SNP genotypes and the proportion of patients with no nausea
The proportion of patients achieving total control in the overall stage, the early stage (0 to 24 hours), and the delayed stage (25 to 120 hours). | 120 hours
  The proportion of patients achieving overall stage, early stage and delayed stage total control is defined as patients who have no vomiting/retching or rescue medications, and no nausea, specifically indicated by a nausea Visual Analog Scale score of 0 during 0 to 120 hours, 0 to 24 hours, and 25 to 120 hours after the initiation of chemotherapy, respectively
The proportion of patients achieving complete protection in the overall stage, the early stage (0 to 24 hours), and the delayed stage (25 to 120 hours) | 120 hours
  The proportion of patients achieving overall stage, early stage and delayed stage complete protection is defined as patients who have no vomiting/retching or rescue medications, and no significant nausea, specifically indicated by a nausea Visual Analog Scale score of less than 25 mm during 0 to 120 hours, 0 to 24 hours, and 25 to 120 hours after the initiation of chemotherapy, respectively
The proportion of no significant nausea in the overall stage, the early stage (0 to 24 hours), and the delayed stage (25 to 120 hours) | 120 hours
  The proportion of patients achieving overall stage, early stage and delayed stage no significant nausea is defined as patients who have no significant nausea, specifically indicated by a nausea Visual Analog Scale score of less than 25 mm during 0 to 120 hours, 0 to 24 hours, and 25 to 120 hours after the initiation of chemotherapy, respectively
The proportion of no nausea (Visual Analog Scale score < 5) in the overall stage, the early stage (0 to 24 hours), and the delayed stage (25 to 120 hours) | 120 hours
  The proportion of patients achieving overall stage, early stage and delayed stage no nausea (Visual Analog Scale score < 5) is defined as patients who have no nausea (Visual Analog Scale score < 5), specifically indicated by a nausea Visual Analog Scale score < 5 mm during 0 to 120 hours, 0 to 24 hours, and 25 to 120 hours after the initiation of chemotherapy, respectively
The proportion of patients achieving complete response in the overall stage, the early stage (0 to 24 hours), and the delayed stage (25 to 120 hours) | 120 hours
  The proportion of patients achieving overall stage complete response is defined as patients who have no vomiting/retching or rescue medications during 0 to 120 hours, 0 to 24 hours, and 25 to 120 hours after the initiation of chemotherapy, respectively
Quality of life in the overall stage | 120 hours
  EuroQol Five Dimensions Questionnaire (EQ-5D) is a standardized instrument used for assessing an individual's health-related quality of life. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has three levels that describe the person's level of functioning or well-being in that specific area. Additionally, EQ-5D includes a Visual Analog Scale where individuals rate their overall health on a scale from 0 (worst imaginable health) to 100 (best imaginable health)
Insomnia | 120 hours
  The proportion of patients with insomnia evaluated by Common Terminology Criteria for adverse events Version 5.0 during 0 to120 hours after the initiation of chemotherapy
Fatigue | 120 hours
  The proportion of patients with fatigue evaluated by Common Terminology Criteria for adverse events Version 5.0 during 0 to120 hours after the initiation of chemotherapy
Constipation | 120 hours
  The proportion of patients with constipation evaluated by Common Terminology Criteria for adverse events Version 4.0 during 0 to120 hours after the initiation of chemotherapy
The side effects of electroacupuncture treatment | 120 hours
  The proportion of side effects related to electroacupuncture treatment in patients evaluated by Common Terminology Criteria for adverse events Version 5.0 during 0 to120 hours after the initiation of chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Qinghai University Affiliated Hospital, Xining, Qinghai, China